CLINICAL TRIAL: NCT04150549
Title: Fecal Microbial Transplantation for Relapsing Multiple Sclerosis Patients - a Placebo-controlled, Double-blinded, Randomized Trial
Brief Title: FMT for MS Patients
Acronym: MS-FMT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Michael Silverman, MD, Chair/Chief of Infectious Diseases, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MS-FMT 002
Record Dates: First submitted 2019-10-11; First posted 2019-11-04 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Transplants (Placebo Comparator)
  Interventions: Biological: Fecal Microbial Transplants
- Allogeneic Transplants (Active Comparator)
  Interventions: Biological: Fecal Microbial Transplants

INTERVENTIONS:
Biological: Fecal Microbial Transplants — Healthy donor stool will be processed and placed into capsules.
  Arms: Allogeneic Transplants
Biological: Fecal Microbial Transplants — Participants stool will be processed and placed into capsules.
  Arms: Autologous Transplants

SUMMARY:
This is a placebo-controlled, double-blinded, randomized trial design, whereby all patients are eligible to start an injectable therapy, and then randomized to either placebo or FMT for approximately 1 year.

DETAILED DESCRIPTION:
Fecal Microbiome Transplants: Patients will undergo pretreatment with Amoxicillin/Clavulinate (or matched placebo) for 5 days followed by a bowel cleanse with PEGLYTE. Patients will undergo allogeneic or autologous fecal transplants. Patients will be dosed with FMT oral capsules approximately 48 hours after antibiotic treatment has stopped. Following the FMT capsule treatment on day 1, patients will be administered a repeat oral capsule or placebo dose at 3 weeks. Oral omeprazole or omeprazole placebo will be given 1 hour prior to the baseline and 3 week dose. This will be done to ensure full engraftment of the transplant.

Participants will be seen at baseline, 3 weeks, 6 weeks, 3 months, 6 months and 12 months. A series of neurological tests will be performed for safety measures. In addition to this, MRIs will be completed at baseline, 6 weeks and 12 months. Blood, urine and stool samples will also be collected for data analysis and safety measures.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 55 years of age
* Have an expanded disability status scale (EDSS) of < 6
* Have a diagnosis of relapsing multiple sclerosis
* Have evidence of radiographic activity within the 12 months on MRI (new/enlarging T2 lesion or gadolinium enhancing lesion)
* Eligible to start/starting an injectable DMT
* Not on a DMT currently and/or not on a DMT in last 6 months
* Ability to swallow capsules

Exclusion Criteria:

* Unable to provide informed consent
* Does not pass the standard MRI screening questionnaire
* Other disease that can affect GI permeability (such as Inflammatory Bowel Disease, Crohn's disease, ulcerative colitis, indeterminate colitis or microscopic colitis, celiac disease)
* Expected requirement for antibiotics within 3 months (chronic suppressive therapies, elective prosthetic joint insertion)
* Toxic megacolon, small bowel ileus
* Penicillin allergy
* Omeprazole allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Changes in T2 Lesions - MRI | Baseline, 6 weeks, 12 months
  Assess the number of new/enlarging/gad enhancing T2 lesions. We will be comparing baseline to 6 weeks and 6 weeks to 12 months.

SECONDARY OUTCOMES:
Blood Brain Barrier - MRI | Baseline, 6 weeks, 12 months
  We will assess the integrity of the blood brain barrier through MRI from baseline to 6 weeks and 6 weeks to 12 months.
Neurofilament Light Serum Levels | Baseline, 6 weeks, 3 months, 12 months
  As a biomarker of neuronal damage neurofilament light chain levels will be detected. Peripheral blood will be collected in appropriate tubes at baseline, 6 weeks, 3 months and 12 months and processed for serum.
  Once collected all samples will be sent to the University of Ottawa where a Simoa NfL assay will be undertaken on their Simoa Analyzer.
  Patients with multiple sclerosis have been shown to have increased intestinal permeability, likely due to a reduction in butyrate-producing bacteria. A decrease in butyrate producing bacteria has been shown to be associated with increased intestinal permeability. Relapsing-remitting MS patients have been shown to have increased intestinal permeability, which may allow dietary and microbial antigens from the intestinal lumen to pass into the blood stream and cause autoimmune responses in MS patients. This may prime the immune system to develop a humoral response to certain bacteria.
Intestinal Permeability | Baseline, 6 weeks, 12 months
  Small Intestine Permeability: Mannitol/Lactulose administration will be used and urine will be collected to measure small intestine permeability. For small intestine permeability patients will be instructed to drink lactulose solution and collect the urine throughout the night and first thing in the morning. A proper collecting bottle will be provided. Once the urine sample bottle reaches the laboratory University Hospital the total volume will be measured and an aliquot of 30mL total, 10mL in each sterile urine container (no other additives) will be separated and stored at -20C and sent on dry ice to Dr. Meddings laboratory at Calgary, Alberta. All biological material will be transported according to biosafety regulations.
IgA Microbiota | Baseline, 3 weeks, 6 weeks, and 12 months
  IgA Microbiota analysis: IgA bound bacteria will be detected and sorted (magnetic beads or flow cytometry) using anti-IgA (pan-IgA, detect monomer and secreted multimer (Miltenyi clone: IS11-8E10). Sorted IgA bound bacteria will be stored, and the DNA extracted in one batch at the end of the study. Changes in the composition of IgA bound bacteria for each patient will be determined using the previously mentioned methods. (Rojas, et al. 2018; Planer, et al. 2016)
Stool Microbiome | Baseline, 3 weeks, 6 weeks, 3 months, 6 months, 12 months
  Gut microbiota analysis before and after FMT: Toilet paper samples will be collected from patients' at baseline and 1-2 days before each scheduled appointment (Al et al. 2018). Patients will store the toilet paper inside of DNA free plastic bags and keep them at 4 °C in the refrigerator until the time of their appointment (alternatively, the samples can be mailed in to the lab, but one method must be chosen for all of the samples collected). Toilet paper samples will be collected from the FMT donor every time they drop off a stool sample for donation. DNA from the toilet paper samples will be extracted in one batch at the end of the study and sent for Illumina Mi-Seq next-generation sequencing of the V4 region of the 16S rRNA gene. Changes in the composition of gut bacteria will be determined using custom R scripts.
Metabolomics | Baseline, 3 weeks, 6 weeks, 3 months, 6 months, 12 months
  Metabolomics: Serum will be collected for metabolomic analysis. Metabolomics can be used to identify biomarkers of MS and may provide us with information about which patients are more likely to respond to FMT therapy. Butyrate producing bacteria have been shown to be in lower relative abundance in MS patients and concentrations of short-chain fatty acids in stool and will be investigated before and after FMT.
Metabolomics | Baseline, 3 weeks, 6 weeks, 3 months, 6 months, 12 months
  Metabolomics: Urine will be collected for metabolomic analysis. Metabolomics can be used to identify biomarkers of MS and may provide us with information about which patients are more likely to respond to FMT therapy. Butyrate producing bacteria have been shown to be in lower relative abundance in MS patients and concentrations of short-chain fatty acids in stool and will be investigated before and after FMT.